CLINICAL TRIAL: NCT04744155
Title: Multi-level Intervention to Reduce Pregnancy Risk Among Adolescents: A Feasibility Trial in the Emergency Department
Brief Title: Reducing Adolescent Pregnancy in the Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Melissa Miller, Study Principal Investigator, Children's Mercy Hospital Kansas City
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY00001169; 1R21HD098086-01A1 (NIH)
Record Dates: First submitted 2020-12-28; First posted 2021-02-08 (Actual); Results first posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Contraception; Adolescent Behavior; Emergency Department
MeSH Terms: conditions — Adolescent Behavior; Emergencies

STUDY DESIGN:
Intervention Model Description: Adolescents will be enrolled into one of two arms: The Multi-level intervention (MLI) or Enhanced Standard of Care (eSOC). Adolescents in both arms will receive motivational interviewing enhanced counseling and a referral for follow up care. Those randomized in the MLI arm will be offered immediate ED-based contraception in addition to receiving a warm referral (providing help with scheduling follow-up care)
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessor will not be aware.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Multi-Level Intervention (Experimental): All adolescents receive the Motivational Interviewing (MI) enhanced counseling and clinic referral.Those randomized to MLI will be offered immediate, ED-based contraception (i.e., oral pill, transdermal patch, vaginal ring, injection, subdermal implant) in addition to receive a warm referral (provider helping to schedule follow-up appointment) to follow-up on selected method (or to initiate in clinic, if preferred)
  Interventions: Behavioral: Multi-Level Intervention
- Enhanced Standard of Care (Active Comparator): All adolescents receive the Motivational Interviewing (MI) enhanced counseling and clinic referral. eSOC participants may obtain contraception only at the referral.
  Interventions: Behavioral: Enhanced Standard of Care

INTERVENTIONS:
Behavioral: Multi-Level Intervention — Behavioral intervention that assesses uptake of contraception and seeks follow-up care.
  Arms: Multi-Level Intervention
Behavioral: Enhanced Standard of Care — Behavioral intervention that assesses uptake of contraception from follow-up care.
  Arms: Enhanced Standard of Care

SUMMARY:
A multi-site randomized trial. Adolescents enrolled in this Clinical Trial will be enrolled into one of two arms. Adolescents in both arms will receive motivational interviewing enhanced counseling and a referral for follow up care. Those randomized in the Multi-level intervention arm will be offered immediate Emergency Department based contraception in addition to receiving a warm referral (providing help with scheduling follow-up care).

DETAILED DESCRIPTION:
Unintended adolescent pregnancy is a major public health problem linked to pregnancy-induced hypertension, low birthweight, and prematurity. In addition, adolescent pregnancies cost an estimated $9.4 billion annually. Though declining, U.S. rates remain among the highest in the developed world. Highly effective methods exist, but adolescents face unique, multi-level barriers to contraceptive access and use. Thus, the vast majority of pregnancies are due to contraceptive non-use or incorrect use. Many, especially minority and uninsured youth, do not attend health maintenance visits; among those who do, seconds is spent discussing sexuality and contraceptive use is not routinely assessed. Multi-level interventions to increase access to contraceptive counseling and all contraceptive types are desperately needed.

As adolescent access to affordable, confidential contraceptive care has worsened in recent years, one approach to increase access is to utilize non-traditional settings, such as Emergency Departments (EDs). The Society for Academic Medicine recognizes the ED as an "effective site for preventive care," evidenced by organizational conferences, consensus statements, and specialized training opportunities to reduce disparities stemming from social determinants of health. Adolescents make 19 million ED visits annually, commonly for non-urgent or reproductive complaints; for many, this may be their only contact with a provider. Adolescents in the ED frequently report unprotected intercourse. The pregnancy risk index (PRI), an estimate of pregnancy risk in the subsequent 12 months, for adolescent females in two EDs was more than three times greater than the national average. Lacking a primary provider was associated with higher PRI scores. While the need for reproductive care is evident, the majority of ED-based studies have focused on screening for sexually transmitted infections (STIs) including HIV and a few, primarily single-site studies have reported on acceptability of hypothetical reproductive care. Among the few addressing pregnancy prevention, most focused on emergency contraception or increasing clinic referral, with mixed results. A small open trial provided counseling and clinic referral for those wanting to initiate contraception. Only 22% completed the referral and one was found to be pregnant at her first clinic visit. Lack of transportation was the most common reason for not completing referral. Because interventions to address multi-level barriers and increase contraception access are sorely needed, the investigator aims to evaluate the feasibility of a novel ED-based intervention, utilizing a mixed methods approach.

Scientific Premise: Many adolescents in the ED are at high-risk of pregnancy yet accepting of reproductive intervention; however, no work describes best practices for ED-based contraceptive provision. Thus, the investigator proposes a randomized trial to evaluate MLI, which includes ED-based contraceptive initiation (i.e., oral pill, transdermal patch, vaginal ring, injection, or subdermal implant) vs. eSOC, for adolescents in two EDs utilizing APPs in a collaborative care model. Thus, the investigator will use a rigorous framework from Bowen et al. to evaluate feasibility constructs (see Table 1 for construct definitions) among adolescents and organizational personnel (i.e., study Advanced Practice Practitioners (APPs), adolescent medicine specialists, ED nursing and Reducing Adolescent Pregnancy in the Emergency Department leaders) in two unique EDs.

ELIGIBILITY:
Inclusion Criteria:

* Females who report past/anticipated intercourse with a male partner within previous year or intent to be sexually active with a male partner in next few months
* Do not desire pregnancy
* Not using intrauterine device (IUD) or Sub-dermal Implant
* English-speaking

Exclusion Criteria:

* Females who report current pregnancy or have positive urine pregnancy test
* Patient has a developmental delay limiting participation
* Patient is presenting in the ED after sexual assault
* Patient is too ill to be screened

Ages: 15 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 37 (Actual)
Dates: Start 2021-05-12 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2023-05-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Children's Mercy Hospital, Kansas City, Missouri
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Study information will be shared with other members on the research team. Study data will be collected and stored via the Research Electronic Data Capture (REDCap) system. De-identifiable information may also be shared with other researchers.
Supporting Information: SAP

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Multi-Level Intervention | Enhanced Standard of Care
Started | 25 | 12
Completed | 25 | 10
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Multi-Level Intervention | Enhanced Standard of Care | Total
Number analyzed (Participants) | 25 | 12 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.5 (0.9) | 16.7 (1.0) | 16.6 (1.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 12 | 37
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 7
  Not Hispanic or Latino | 21 | 9 | 30
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 19 | 8 | 27
  White | 3 | 0 | 3
  other | 3 | 4 | 7
Previous sexual activity [Number; unit: participants] | 15 | 9 | 24
Previous hormonal contraception use [Count of Participants; unit: Participants] | 11 | 7 | 18

OUTCOME MEASURES:

1. Primary Outcome: Adolescent Feasibility of Intervention
Description: The intervention will be deemed feasible if the median score across all items is ≥ 3. Individual responses range from 1 to 5. Higher scores indicate greater feasibility using the investigator created Feasibility Assessment.
Time Frame: 1 visit on day 1
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Groups:
- Multi-level Intervention: Adolescent participants who received the counseling intervention and opportunity to start contraception at index visit
- Enhanced Standard of Care: Received counseling but no opportunity for same day initiation, they received referral only.
Arm/Group | Multi-level Intervention | Enhanced Standard of Care
Number analyzed (Participants) | 16 | 9
score on a scale | 4.5 [4.2 to 4.8] | 4.7 [4.6 to 5.0]

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- Enhanced Standard of Care: Adolescent participants who received the eSOC intervention
- Multi-level Intervention: Adolescent participants who received the MLI intervention
Arm/Group | Enhanced Standard of Care | Multi-level Intervention
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/25
Other Adverse Events (participants affected / at risk) | 0/12 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2022-04-12): https://cdn.clinicaltrials.gov/large-docs/55/NCT04744155/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-19): https://cdn.clinicaltrials.gov/large-docs/55/NCT04744155/SAP_001.pdf
  • Informed Consent Form (2022-02-09): https://cdn.clinicaltrials.gov/large-docs/55/NCT04744155/ICF_002.pdf